CLINICAL TRIAL: NCT05299190
Title: Feasibility, Acceptability and Preliminary Efficacy of a Hospital-based Antenatal Yoga Program for Anxious and Depressed Women
Brief Title: Antenatal Yoga Intervention for Depressed and Anxious Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment challenges due to COVID-19 pandemic
Sponsor: Hopital Montfort (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HMontfort
Record Dates: First submitted 2020-02-26; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2019-08

CONDITIONS: Anxiety Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the yoga intervention plus treatment as usual (TAU) or TAU plus biweekly clinical monitoring
Who Masked: Outcomes Assessor
Masking Description: The MINI will be administered at 6-months post-partum by a blind assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga intervention plus TAU (Experimental): Participants randomized to the yoga intervention will attend 8-weekly 90-minute group sessions. The intervention will be delivered by certified instructors with experience facilitating yoga classes for pregnant women. Monthly "drop-in" classes will be scheduled in order to motivate women to maintain their practice during the follow-up period. The yoga intervention will be based on the hatha yoga system modified for pregnancy. TAU will include treatment based on the recommendation of participants' healthcare provider/team.
  Interventions: Other: Yoga intervention plus TAU
- Clinical Monitoring plus TAU (Other): Clinical monitoring will be conducted by telephone and include a 15-20 minutes discussions of how the participant has been feeling over the past two weeks. A standard format will be used for conducting the clinical monitoring telephone calls. TAU will include treatment based on the recommendation of participants' healthcare provider/team.
  Interventions: Other: Clinical Monitoring plus TAU

INTERVENTIONS:
Other: Yoga intervention plus TAU — The yoga intervention consists of 8 weekly group sessions. The intervention is based on hatha yoga system. TAU is usual care participants receive from their health care provider
  Arms: Yoga intervention plus TAU
Other: Clinical Monitoring plus TAU — clinical monitoring includes bi-weekly 15-20 minute telephone contact with participants. TAU is usual care participants receive from their health care provider.
  Arms: Clinical Monitoring plus TAU

SUMMARY:
The aim of this study is to determine if a hospital-based antenatal yoga program (HB-AYP) is a feasible, acceptable and potentially efficacious intervention for women with antenatal anxiety and/or depression?

DETAILED DESCRIPTION:
Anxiety and depression are the most common psychological symptoms reported in pregnant women and can result in adverse obstetric, neonatal and post-partum mental health outcomes. Although there is a range of effective first-line treatments for anxiety and depression, these treatments are not without limitations. Concerns about the safety of antidepressant medication during pregnancy, lack of access to affordable psychosocial treatments and reluctance to seek mental health care due to stigma may prevent pregnant women from receiving optimal care for their symptoms. Recently, there has been growing interest in alternative and complementary approaches to manage anxiety and depression. These approaches may offer women with antenatal anxiety and depression an alternative treatment option that may be more acceptable and perceived as more holistic and less stigmatizing than conventional mental health care. One way to optimize access to yoga therapy during prenatal care is to implement an antenatal yoga program within a public healthcare system. Accordingly, the overarching aim of this study is to evaluate the feasibility of a hospital-based antenatal yoga program (HB-AYP) plus treatment as usual for anxiety and depression, and obtain preliminary data on its potential efficacy relative to treatment as usual plus biweekly clinical monitoring(TAU) This pilot research will provide much needed preliminary data that will set the foundation for designing a fully-powered prospective randomized controlled trial (RCT) of a HB-AYP. In the long term, it is hoped that this line of research will influence evidence-based clinical guidelines for managing antenatal anxiety and depression and service delivery.

ELIGIBILITY:
Inclusion Criteria: Healthy women in their second trimester of an uncomplicated pregnancy with elevated levels of anxiety and/or depression (based on the PHQ-9 and GAD-7) will be eligible to participate

-

Exclusion Criteria: i) a lifetime history of psychosis, ii) symptoms of mania/hypomania in the past 12 months; iii) a history of substance use disorders in the last 6 months; iv) a history of self-harm in the last 6 months; v) high suicide risk; vi) engaged in a regular formal meditative practice at least once a month over the past 12 months; and vii) yoga postures are contraindicated.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-08-24 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale | Baseline; week 4; week 8; bimonthly until 6 months postpartium
  measure of depressive symptoms

SECONDARY OUTCOMES:
Perceived Stress Scale | Baseline; Week 8; bimonthly until 6-months postpartum;
  measure of stress
Interpersonal Relationships Inventory (interpersonal support subscale) | Baseline; Week 8; 6-months post-partum
  Measure of interpersonal support
Dyadic Adjustment Scale | Baseline; Week 8; 6-months post-partum
  Measure of marital adjustment
Five Facet Mindfulness Scale | Baseline; Week 8; 6-months post-partum
  Measure of facets of mindfulness
Self-Compassion Scale | Baseline; Week 8; 6-months post-partum
  Measure of self-compassion
Prenatal Attachment Inventory | Baseline; Week 8
  Measure of prenatal attachment
Post-partum bonding questionnaire | 6-months postpartum
  Measure of post-partum bonding

OTHER OUTCOMES:
Feasibility outcomes | Week 1 to 8
  Ease of recruitment; study compliance, program satisfaction; perception of treatment credibility
Pregnancy outcomes | Baseline and week 8 and post-partum
  Presence of gestational diabetes and hypertension; gestational age at delivery, mode of delivery, pregnancy and birth complications, infant birth weight; Apgar scores
Stress hormones | Baseline and week 8 for mother and 8-weeks and 6-months for infant
  Salivary cortisol and alpha amylase

CONTACTS AND LOCATIONS:
Overall Officials: Diana Koszycki, PhD, Principal Investigator — Institut du Savoir Montfort

IPD SHARING:
Plan to Share IPD: No